CLINICAL TRIAL: NCT04511585
Title: The "Great Live and Move Challenge": a Program to Promote Physical Activity Among Children Aged 7-11 Years. Design and Implementation of a Cluster-randomized Controlled Trial.
Brief Title: The "Great Live and Move Challenge" Among Children Aged 7-11 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Collaborators: Laboratoire EPSYLON (Unknown); Academic resource center of herault (Unknown); University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EPIDAURE- 2017/01
Record Dates: First submitted 2017-08-28; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: a 24-month (6 weeks each year) multilevel and TPB-based program aiming to promote PA practice
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLMC experimental arm (Experimental): GLMC experimental arm receiving a 24-month (6 weeks each year) multilevel and TPB-based program aiming to promote PA practice
  Interventions: Behavioral: Great Live and Move Challenge
- the control arm (No Intervention): the control arm that do not receive any intervention

INTERVENTIONS:
Behavioral: Great Live and Move Challenge — Physical activity program for children
  Arms: GLMC experimental arm

SUMMARY:
The Great Live and Move Challenge (GLMC) study is a 2-year cluster-randomized controlled trial designed to evaluate a multilevel and theory-based intervention to promote PA practice in children aged 7-11 years from French primary schools.

DETAILED DESCRIPTION:
Recent population-based surveys have reported that a large majority of children were not active enough to meet the physical activity (PA) international guidelines in France, Europe and in the US. Therefore, there is a need to find efficient programs to improve PA habits in children from early age. The Great Live and Move Challenge (GLMC) study is a 2-year cluster-randomized controlled trial designed to evaluate a multilevel and theory-based intervention to promote PA practice in children aged 7-11 years from French primary schools. The aim of this paper is to describe the GLMC study protocol. The primary hypothesis is that the GLMC intervention will increase by 15% the proportion of children meeting the World Health Organization recommendations of 60 minutes/day of moderate to vigorous PA. Study recruitment goal is 5000 children . The GLMC is implemented on children and their parents and involves multiple local grass-roots partners, such as school teachers and municipal officials, as well as policy stakeholders. The Theory of Planned Behavior (TPB) constitutes the foundations of the intervention conception. The total duration of the intervention is 3.5 months each year, for two years. Children and parents are evaluated at pre- and post-intervention every year regarding PA practice (self-reported and objectively measured in a subsample of 400 children), TPB variables (i.e., intentions, attitudes, subjective norms, perceived behavioral control) and other psychosocial variables (e.g., perceptions of active opportunities). This study will evaluate the effectiveness of a multilevel and theory-based primary school PA program and potentially provide valuable information for schools and public health policers looking for innovative PA programs.

ELIGIBILITY:
Inclusion Criteria:

* All the children (and their parents) schooled in a primary school (year 3 or year 4) from Hérault, Gard, and Aude French departments

Exclusion Criteria:

* none

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5000 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Physical activity practice in hours per week in children is self-recorded | up to 3.5 years
  physical activity practice in hours per week in children is self-recorded using an adapted version of the self-administered Physical Activity Questionnaire for Children (PAQ-C)

CONTACTS AND LOCATIONS:
Overall Officials: Florence cousson gelie, Principal Investigator — Epidaure, prevention department of ICM
Locations (1):
- Institut régional di Cancer de Montpellier (ICM), Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided